CLINICAL TRIAL: NCT01675713
Title: Intensive Lifestyleintervention for the Treatment of Severe Obesity
Brief Title: Lifestyleintervention for the Treatment of Severe Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Hjelp24 (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, PhD, Norwegian School of Sport Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KKD1
Record Dates: First submitted 2012-08-20; First posted 2012-08-30 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Morbid Obesity
Keywords: Lifestyle; Physical activity
MeSH Terms: conditions — Obesity, Morbid; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle intervention (Experimental): 10-14 weeks intensive lifestyle intervention
  Interventions: Behavioral: Intensive lifestyle intervention
- Controls (No Intervention): No treatment, waiting list

INTERVENTIONS:
Behavioral: Intensive lifestyle intervention — Lifestyle modification program focusing on increasing physical activity level, adjusting energy intake and learning coping strategies
  Arms: Lifestyle intervention

SUMMARY:
The overall purpose of this project is to study the acute, short- (≤ 1 year) and long- (> 1 year) term effects on body composition and psychological health after a 10 to 14-weeks comprehensive lifestyle modification program for the treatment of severe obesity.

The aims of the PhD project are to investigate whether an intensive lifestyle intervention leads to acute and short term (< 1 year) changes in:

1. The BMI/Weight
2. Body composition (waist circumference, fat mass, fat free mass, skeletal muscle mass and visceral fat area)
3. Psychosocial factors such as eating behavior, anxiety and depression symptoms and health-related quality of life

DETAILED DESCRIPTION:
The study is based on data collected from patients at The Hjelp24 NIMI Ringerike Obesity Clinic, which is an inpatient program to address morbid obesity in adults. The study is a non-randomized clinical trial comparing the acute and long-term effects on physical and psychological health of the 10-14-weeks inpatient comprehensive lifestyle modification program for the treatment of morbidly obese patients.

In between the inpatient stay, the patients are followed up either by telephone, occasional mail and/or structured / weekly email.

In this project we prospectively follow two groups of patient included in the treatment programme in September 2010 and January 2011, respectively. In addition a control group with waiting-list patients is also included in the study, and they were recruited in October-November 2011

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese

Exclusion Criteria:

* not able to walk slowly for 20 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Acute and short term (12 months) effects of an intensive 10 to 14-weeks inpatient program with lifestyle modification for the treatment of morbidly obese patients on body composition and psychosocial health | three years

SECONDARY OUTCOMES:
Body composition | Week 10-14
  Change in body composition (body weight, fat mass, fat free mass, visceral fat area) from baseline
Body composition | Week 26
  Change in body composition (body weight, fat mass, fat free mass, visceral fat area) from baseline
Body composition | Week 52
  Change in body composition (body weight, fat mass, fat free mass, visceral fat area) from baseline
Health related quality of life | Week 10-14
  Change in Health related quality of life from baseline
Health related quality of life | Week 26
  Change in Health related quality of life from baseline
Health related quality of life | Week 52
  Change in Health related quality of life from baseline
Binge Eating | Week 10-14
  Change in binge eating from baseline
Binge eating | Week 26
  Change in binge eating from baseline
Binge eating | Week 52
  Change in binge eating from baseline
Anxiety | Week 10-14
  Change in anxiety from baseline
Depression | Week 10-14
  Change in depression from baseline
Depression | Week 26
  Change in depression from baseline
Depression | Week 52
  Change in depression from baseline
Physical Activity | Week 10-14
  Change in physical activity from baseline
Physical activity | Week 26
  Change in physical activity from baseline
Physical activity | Week 52
  Change in physical activity from baseline
Physical fitness | Week 10-14
  Change in physical fitness from baseline
Physical fitness | Week 26
  Change in physical fitness from baseline
Physical fitness | Week 52
  Change in physical fitness from baseline
Systolic Blood Pressure | Week 10-14
  Change in Systolic Blood Pressure
Systolic Blood Pressure | Week 26
  Change in Systolic Blood Pressure
Systolic Blood Pressure | Week 52
  Change in Systolic Blood Pressure from baseline
Lipids | Week 10-14
  Change in lipids (Total cholestrol, LDL cholestrol, HDL cholestrol and Triglycerides) from baseline
Lipids | Week 26
  Change in lipids (Total cholestrol, LDL cholestrol, HDL cholestrol and Triglycerides) from baseline
Lipids | Week 52
  Change in lipids (Total cholestrol, LDL cholestrol, HDL cholestrol and Triglycerides) from baseline
Glucose | Week 10-14
  Change in glucose from baseline
Glucose | Week 26
  Change in glucose from baseline
Glucose | Week 52
  Change in glucose from baseline
Explore the participants experiences with physical activity prior to, during and after the treatment programme | 2-3 years post treatment
  In depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Mæhlum, MD, PhD, Study Director — Hjelp24
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

REFERENCES:
- [Background] Maehlum S, Danielsen KK, Heggebo LK, Schioll J. The Hjelp24 NIMI Ringerike obesity clinic: an inpatient programme to address morbid obesity in adults. Br J Sports Med. 2012 Feb;46(2):91-4. doi: 10.1136/bjsm.2010.071894. Epub 2010 May 10. PMID 20460258
- [Result] Danielsen KK, Sundgot-Borgen J, Maehlum S, Svendsen M. Beyond weight reduction: improvements in quality of life after an intensive lifestyle intervention in subjects with severe obesity. Ann Med. 2014 Aug;46(5):273-82. doi: 10.3109/07853890.2013.874660. Epub 2014 Feb 4. PMID 24491067
- [Result] Danielsen KK, Svendsen M, Maehlum S, Sundgot-Borgen J. Changes in body composition, cardiovascular disease risk factors, and eating behavior after an intensive lifestyle intervention with high volume of physical activity in severely obese subjects: a prospective clinical controlled trial. J Obes. 2013;2013:325464. doi: 10.1155/2013/325464. Epub 2013 Apr 22. PMID 23710347